CLINICAL TRIAL: NCT06532149
Title: ERectile Dysfunctions, gOnadotoxicity and Sexual Health Assessment in Men With Lung Cancer (EROS)
Brief Title: ERectile Dysfunctions, gOnadotoxicity and Sexual Health Assessment in Men With Lung Cancer
Acronym: EROS
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Bria Emilio, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6578
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: NSCLC Stage IV; Sex Disorder; Hypogonadism, Male; Erectile Dysfunction
Keywords: NSCLC; Sexual Health; Male hypogonadism; Erectile Dysfunction
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Sexual Dysfunction, Physiological; Eunuchism; Erectile Dysfunction | interventions — alectinib; brigatinib; lorlatinib; osimertinib; sotorasib; dabrafenib; trametinib; selpercatinib; pembrolizumab; cemiplimab; Nivolumab; Carboplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma sample for full hormone assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A: Male patients diagnosed with advanced/metastatic ALK+ o ROS-1+ NSCLC, who are receving active anticancer treatment
  Interventions: Drug: Alectinib; Drug: Brigatinib; Drug: Lorlatinib 100 mg
- Cohort B: Male patients diagnosed with advanced/metastatic oncogene-addicted NSCLC (other than ALK and ROS-1), who are receving active anticancer treatment
  Interventions: Drug: Osimertinib; Drug: Sotorasib; Drug: Dabrafenib; Drug: Trametinib; Drug: Selpercatinib
- Cohort C: Male patients diagnosed with advanced/metastatic non oncogene-addicted NSCLC, who are receving immunotherapy (single agent or combintions without cytotoxic agents)
  Interventions: Drug: Pembrolizumab; Drug: Cemiplimab; Drug: Nivolumab
- Cohort D: Male patients diagnosed with advanced/metastatic non oncogene-addicted NSCLC, who are receving chemotherapy alone or in combination with immunotherapy
  Interventions: Drug: Pembrolizumab; Drug: Cemiplimab; Drug: Nivolumab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel

INTERVENTIONS:
Drug: Alectinib — Alectinib 600 mg/BID
  Other Names: Alecensa
  Groups: Cohort A
Drug: Brigatinib — 180 mg/daily
  Other Names: ALUNBRIG
  Groups: Cohort A
Drug: Lorlatinib 100 mg — 100 mg/daily
  Other Names: LORVIQUA
  Groups: Cohort A
Drug: Osimertinib — 80 mg/daily
  Groups: Cohort B
Drug: Sotorasib — 960 mg/daily
  Groups: Cohort B
Drug: Dabrafenib — 150 mg/BID
  Groups: Cohort B
Drug: Trametinib — 2 mg/daily
  Groups: Cohort B
Drug: Selpercatinib — 160 mg/BID
  Groups: Cohort B
Drug: Pembrolizumab — 200 mg intravenous every 21 days
  Groups: Cohort C; Cohort D
Drug: Cemiplimab — 350 mg intravenous every 21 days
  Groups: Cohort C; Cohort D
Drug: Nivolumab — 240 mg intravenous every 14 days
  Groups: Cohort C; Cohort D
Drug: Carboplatin — AUC4/AU5 intravenous every 21 days
  Groups: Cohort D
Drug: Pemetrexed — 500 mg/mq intravenous every 21 days
  Groups: Cohort D
Drug: Paclitaxel — 175 mg/mq intravenous every 21 days
  Groups: Cohort D

SUMMARY:
Although many phase III clinical trials evaluate the quality of life as a secondary endpoint, male sexuality remains a neglected topic in oncology research. In light of the long-term efficacy of new-generation anticancer treatments for ANSCLC (i.e. targeted therapies and immunotherapy), there is a paucity of data about any detrimental effect on fertility and sexuality that could complicate the therapy proposal, especially in young patients.

The aim of this trial is to assess incidence of endocrine toxicity and sexual dysfuction in male patients receiving active treatment for ANSCLC

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced/metastatic NSCLC
* To be candidate to active treatment
* Aged ≥ 18 anni (up to 75 years old)
* To be sexually active in last 30 days before treatment start
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Written informed consent

Exclusion Criteria:

* History of endocrine disorders, excepting for controlled hypothyroidism (surgical or non-surgical) treated with replacement levothyroxine since at least 2 years
* Any cancer-related or medical condition that would interfere with the patient reported outcomes or laboratory assessment. Examples include, but are not limited to:
* Cancer-related conditions that may preclude/undermine sexual activity (e.g. leptomeningeal carcinomatosis, pathological vertebral fractures, gonadic metastases, unstable spinal cord compression, uncontrolled neurological symptoms, surgical complications):

  * History of chronic liver disease or hormonal replacement therapy (e.g. ADT for prostatic cancer)
  * Participants who not adequately recovered from previous confirmed chemotherapy-induced gonadotoxicity (e.g. cisplatin)
  * Chronic use of drugs with known effect on male sexuality, including opiates, anxiolytics, antidepressants, mood stabilizers, beta blockers (e.g. atenolol) and high dose diuretics
  * Psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
  * Major psychological disorder and/or high distress level that would interfere with sexual function and the participant's ability to cooperate with the requirements of the study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sexually active male patients diagnosed with advanced/metastatic NSCLC who are receiving active treatement according to their tumor molecular profiling
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related sexual dysfuction in male patients with ANSCLC | From treatment start up to 1 year
  Percentage of patients who reported any sexual health disorders after treatment start

SECONDARY OUTCOMES:
Incidence of treatment-related hypogonadism in male patients with ANSCLC | From treatment start up to 1 year
  Percentage of patients who reported reduction of testosterone levels after treatment start
Incidence of treatment-related erectile dysfuction in male patients with ANSCLC | From treatment start up to 1 year
  Percentage of patients who erectile dysfuction after treatment start

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No